CLINICAL TRIAL: NCT00328432
Title: Phase IB Study of Biomarker Modulation by Celecoxib vs. Placebo in Women With Newly-Diagnosed Breast Cancer
Brief Title: A Study of Women With an Early Diagnosis of Breast Cancer, Taking Celecoxib Between the Biopsy and Lumpectomy/Mastectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Kansas (Other)
Collaborators: Pfizer (Industry)
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 9061
Record Dates: First submitted 2006-05-19; First posted 2006-05-22 (Estimated); Last update posted 2008-09-17 (Estimated); Status verified 2008-09

CONDITIONS: Breast Cancer
Keywords: early breast cancer; double-blind randomized placebo-controlled; RCT; pre-surgical model; DCIS model; COX-2 inhibitor; celecoxib; Ki-67 placebo
MeSH Terms: conditions — Breast Neoplasms | interventions — Celecoxib; BID protein, human

INTERVENTIONS:
Drug: celecoxib 400 mg bid

SUMMARY:
To assess the effects of short term administration of celecoxib 400 mg bid between biopsy and reexcision.

DETAILED DESCRIPTION:
A double blind randomized study of celecoxib 400 mg bid versus placebo in newly diagnosed breast cancer. Assessment of modulation of tissue markers (Ki-67, ER, VEGF, PR, etc.) and serum markers (estradiol, estrone, SHBG, etc.).

ELIGIBILITY:
Inclusion Criteria:

* women with a recent diagnosis of T1 or T2 non-invasive breast cancer by large core needle or excisional biopsy
* confirmation that tissue was processed in methods acceptable to protocol and sufficient tissue remains post-diagnostic analyses to perform research assessments
* reexcision planned within 10 days to 6 weeks from study start
* if on prevention tamoxifen or raloxifene, must have begun administration at least six weeks prior to initial biopsy and continue through reexcision

Exclusion Criteria:

* no hormone replacement therapy within the 90 days prior to biopsy
* if on prevention tamoxifen or raloxifene, must have begun administration at least six weeks prior to initial biopsy and continue through reexcision
* no evidence of metastatic malignancy of any kind
* no history of asthma, allergy ASA, NSAIDS, celecoxib or other COX-2 inhibitors for a chronic non-oncological condition with the excision of low dose ASA (160 mg daily) during 4 weeks prior to biopsy and for the duration of the study.
* no celecoxib or rofecoxib use within one month of biopsy
* no history of gastrointestinal ulcer or ulcerative colitis requiring treatment
* no current anticoagulants
* no neoadjuvant antihormone or chemotherapy as treatment following biopsy prior to study entry or concurrently with participation on study
* no aromatase inhibitor in the six months prior to participation
* no concomitant lithium
* no known significant bleeding disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2003-06; Study Completion 2005-12

PRIMARY OUTCOMES:
Proliferation marker (Ki-67) in tissue specimens comparing baseline and post-drug administration specimens.

SECONDARY OUTCOMES:
Baseline and post-administration assessments of MAP kinase, pERK1 and 2, activated pAKT, change in apotosis indicators, and angiogenesis associated proteins, and Her-2/neu.

CONTACTS AND LOCATIONS:
Overall Officials: Carol J Fabian, MD, Principal Investigator — University of Kansas Medical Center
Locations (7):
- United States (7):
  - University of Alabama-Birmingham, Birmingham, Alabama
  - MDDesert Comprehensive Breast Center, Palm Springs, California
  - Loyola University Medical Center, Maywood, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cleveland Clinical Foundation, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - US Oncology, Dallas, Texas